CLINICAL TRIAL: NCT00776763
Title: The Profile of the Growth Factors and Other Mediators of Angiogenesis in the Ocular Fluids in Proliferative Retinopathies (AMD and PDR) Before and After the Intravitreal Administration of Bevacizumab (Avastin) as an Anti-VEGF Blocker
Brief Title: Ocular Growth Factors Profile in Proliferative Retinopathies Before and After Intravitreal Bevacizumab
Acronym: KIA-ProRet
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ophthalmological Association Edelweiss (Other)
Collaborators: University of Cologne (Other)
Responsible Party: NARCISA IANOPOL, Md, PhD, Railway Universitary Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KIA-ProRet
Record Dates: First submitted 2008-10-17; First posted 2008-10-21 (Estimated); Last update posted 2011-07-22 (Estimated); Status verified 2008-10

CONDITIONS: Proliferative Diabetic Retinopathy; Age Related Macular Degeneration
MeSH Terms: conditions — Macular Degeneration | interventions — Bevacizumab

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (1):
- Avastin (Experimental)
  Interventions: Drug: Avastin intravitreal injection

INTERVENTIONS:
Drug: Avastin intravitreal injection — 1,25 mg of Bevacizumab (Avastin) will be intravitreally injected 4 weeks interval in the proliferative retinopathies groups (exudative age related macular degeneration and proliferative diabetic retinopathy)

SUMMARY:
Aims of the trial: Establishing the profile of the growth factors and other mediators of angiogenesis in different ocular fluids (aqueous humour, vitreous gel and ocular liquid in vitrectomized eyes), in the 2 most frequent proliferative retinopathies - diabetic proliferative retinopathy (PDR) and exudative age related macular degeneration (AMD). Following up the dynamic of this profile before and after intravitreal administration of Bevacizumab (Avastin) as an anti-VEGF blocker.

Materials: The research will be conducted on the following categories of patients groups:

* nondiabetic patients without AMD or any other diagnosed proliferative ocular disease (controls)
* patients with age related macular degeneration (AMD groups) before and after intravitreal injections with Avastin
* diabetic patients with different types of diabetic retinopathy, before and after intravitreal Avastin (diabetic groups) Methods: Samples from different ocular fluids will be collected from each group of patients. 10 growth factors and other 10 cytokines will be determined in the ocular fluids samples.

Results: The results from the biochemical measurements will be statistically interpreted in order to obtain conclusions for the clinical practice.

Conclusions: The conclusions of this trial will be used exclusively for research publications and communications, as well as for clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* age over 20 years
* nondiabetic patients requiring cataract surgery or vitrectomy for different posterior segment nonproliferative disorders - controls groups
* diabetic patients asking ophthalmologic treatments for different degrees of decreasing of visual acuity - diabetic groups
* diabetic patients requiring cataract surgery or vitrectomy - diabetic groups
* age related macular degeneration patients asking ophthalmologic treatments for different degrees of decreasing of visual acuity - age related macular degeneration groups
* age related macular degeneration patients requiring cataract surgery or vitrectomy - age related macular degeneration groups

Exclusion Criteria:

* patients under the age of 20 years
* patients that did not accept and signed the informed consent of the trial
* patients that received any anti-VEGF therapy for any proliferative or inflammatory ocular disease
* patients that received any type of intraocular injection with any pharmaceutical agent
* patients with any clinical type of malignancy in their pathologic antecedents
* patients with recent penetrating trauma (less than 1 year old)
* patients operated for different ocular disorders requiring combination with antimetabolites (ex. 5-FU or Mitomycin C with trabeculectomy)
* patients with intraocular inflammations or infections or other pathologies that contraindicate open globe surgery or intraocular injections with anti-VEGF blockers

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2008-10; Primary Completion 2009-10 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Growth Factors and Other Cytokines Measurements | 1 month interval

CONTACTS AND LOCATIONS:
Overall Officials: NARCISA IANOPOL, Researcher, Principal Investigator — Railway Universitary Hospital
Locations (1):
- Railway Universitary Hospital, Iași, Romania